CLINICAL TRIAL: NCT03017105
Title: A Study Comparing the Use of Cross-education of Strength-training for the Non-injured Limb With Traditional Rehabilitation After Conservatively Managed Proximal Humerus Fractures in Adult Patients
Brief Title: Cross-education for Proximal Humerus Fracture Rehabilitation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Logistical difficulties leading to an extremely slow recruitment rate
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Jenna Bardsley, Principle Investigator, Liverpool University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5222
Record Dates: First submitted 2017-01-03; First posted 2017-01-11 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Proximal Humerus Fractures (to be Managed Non-operatively)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Usual rehabilitation: non-operative management of the fracture; will undergo usual physiotherapy rehabilitation for the injured arm
  Interventions: Other: Usual rehabilitation
- Experimental (Experimental): Cross-education of strength-training: non-operative management of the fracture; will undergo usual physiotherapy rehabilitation for the injured arm but will also undergo strength-training for the uninjured arm
  Interventions: Other: Cross-education of strength-training; Other: Usual rehabilitation

INTERVENTIONS:
Other: Cross-education of strength-training — Strength-training exercises using isometric contractions and resistance bands to be performed with the uninjured arm
  Arms: Experimental
Other: Usual rehabilitation — Exercises to improve range of movement, strength and movement control (as standard for non-operatively managed proximal humerus fractures)

SUMMARY:
Proximal humerus fractures (break of the top part of the upper arm bone) are common in older people with poorer bone quality. Often patients do not undergo surgery for these fractures: the bone fragments may be in an acceptable enough position to be able to heal naturally, or the patient may not be well enough medically to undergo an operation. These patients need to wear a sling to immobilise their injured shoulder, however muscles start to weaken quickly when they are unable to be used. This research project will look at whether strength-training the opposite/uninjured limb, known as "cross education", has any effect on preserving the function of the injured/fractured limb. Participants will be randomised into two groups using minimisation, that is to say the groups will have balanced numbers in terms of exact pattern of fracture and gender. One group will receive traditional rehabilitation exercises and treatment by the physiotherapist for their injured limb; the other group will receive the same but in addition will also undergo a strength-training exercise programme for their uninjured limb. Only qualified physiotherapists with experience of treating this patient cohort will be involved. Sessions in the physiotherapy department will last up to 30 minutes each and will comprise of: patient review, exercise progression, and advice giving/question answering; home exercise programmes will be expected to be completed 2-3 times daily and last up to 30 minutes each; number of sessions will be agreed between the participant and treating physiotherapist with treating ending once an agreed, acceptable level of function has been achieved. The Oxford Shoulder Score patient-reported outcome measure will be completed by the participant at 6 and 12 weeks and the European Quality of Life (EuroQoL)-5D-5L at 12 weeks after commencement of treatment.

DETAILED DESCRIPTION:
This study will investigate the use of cross education (ie. strength-training the uninjured limb) as part of the recovery and return to function for skeletally mature, adult patients as measured by the Oxford Shoulder Score after proximal humerus fracture and answer the question:

does the use of a strength-training programme for the non-injured limb affect return to function in adult patients with proximal humerus fractures?

Proximal humerus fractures (break to the top part of the upper arm bone) are common, accounting for 4-6% of all fractures in the older population and almost one-fifth of all fractures sustained after a fall from a standing height in patients with osteoporosis. These fractures can functionally impair the upper limb and so impact on overall quality of life. Some studies show that a number of previously fit and independent patients may not return to independent activity following a proximal humerus fracture and may even be at increased risk for sustaining a subsequent fractured hip/neck of femur. If new rehabilitation approaches can help improve the level of function achieved the morbidity and quality of life of these patients could potentially be improved.

The ageing population of the United Kingdom means the number of patients sustaining these fractures will increase and so increase the cost to the National Health Service and the risk of morbidity/mortality/disability/poor health-related quality of life. Treatment needs to address range of movement (ROM) and muscle strength as well as restoration of function and access to the community as quickly as possible. Effective, timely and cost-efficient management of these patients must be found.

Patients with proximal humerus fractures generally undergo a period of wearing a sling to immobilise the limb/stop them from moving it- especially those being managed without an operation. Different orthopaedic and physiotherapy teams across the UK use different periods of immobilisation, start rehabilitation at different times after injury and use different rehabilitation methods. Only a few randomised controlled trials (RCTs) exist looking into when to start physiotherapy and exactly what physiotherapy to do. Studies are needed to develop treatment and rehabilitation protocols to deliver the best and most cost-effective patient care possible.

Wearing a sling/immobilisation of a limb for as little as one week can cause significant muscle wastage resulting in loss of strength and loss of function. Studies have shown that there is up to 60% reduction in strength after 5-6 weeks immobilisation. This early decline in strength could be due to fewer nerve signals being sent from the brain to the inactive muscles. It has been suggested that this could be prevented by strength-training the uninjured limb, known as "cross-education". The exact mechanisms by which it works are still unknown but it is thought that using cross-education could help maintain messages sent from the brain and so minimise changes in muscle and facilitating quicker recovery. The body works reciprocally in many ways, for example swinging the opposite arm (to the stepping leg) whilst walking. Many studies have already been done that show an improvement/maintenance of strength of an immobilised limb after strength-training the opposite limb but these studies have looked at uninjured patients or at those with lower limb injuries. Research into using the principle of cross-education with upper limb injuries is needed before it can be applied in practice routinely to patients.

The patient will be asked some questions by the Specialist Physiotherapist or Doctor during their fracture clinic appointment to see whether they are eligible to take part in the study. If eligible they will have be provided with a written information sheet and the clinician will explain the study and answer any questions they may have.

Patients will receive a phone call from the primary researcher 24-48 hours after being provided with the study information to answer any further questions they may have and to gauge interest in participation in the trial. If they are keen to be involved the primary researcher will arrange for them to come into the Physiotherapy department to sign a written consent form. At this appointment (which will take place in a clinical office within the department) the primary researcher will then use a computer programme (called Minim) to allocate them into one of the two study groups. If they are allocated into the experimental group the primary researcher will teach them their strengthening exercises for their uninjured limb, and will then arrange their first follow up physiotherapy appointment for within the next 2-3 weeks. Patients allocated to the control group (standard rehabilitation) will be booked their first physiotherapy appointment after signing their consent form. The patient will also be asked to complete some questionnaires about their current level of function/pain/etc.- these are completed by all patients suffering this particular injury regardless of participation in the study.

All participants will have ongoing physiotherapy treatment at as many appointments as are deemed necessary in agreement with themselves and the treating physiotherapist to return to their required level of function. Those in the experimental group will receive a strength-training regime for they uninjured limb in addition to usual rehabilitation for the injured limb. Those in the control group will receive usual rehabilitation for the injured limb. All participants will be required to complete further questionnaires at 6 and 12 weeks after the initial questionnaires were completed (as is the case for all patients receiving physiotherapy at this Trust).

ELIGIBILITY:
Inclusion Criteria:

* Proximal humerus fracture <2 weeks old
* Isolated injury sustained
* After low-energy trauma (i.e. simple fall from standing; high-energy injuries often have concurrent injuries or require surgery)
* For conservative management
* English speaking/understanding (for the duration of the pilot; the full study could be extended to include use of translated information and interpreters)
* Independent living at the time of injury (i.e. not institutionalised, so measure of function is a relevant outcome)

Exclusion Criteria:

* Concurrent injuries
* Fractured shaft of or distal humerus
* Pathological fracture (due to cancer) or fracture as a result of high energy trauma
* Previous fracture or pathology to either side
* History of upper extremity neurological problems (e.g. multiple sclerosis, stroke, Parkinson's disease, vestibular disorders, reflex neuropathy)
* Diagnosis of dementia/other cognitive impairment
* Not able to attend the Trust's outpatient departments for rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 12 weeks after injury

SECONDARY OUTCOMES:
EuroQoL-5D-5L | at 6 weeks & 12 weeks after injury
Oxford Shoulder Score | at 6 weeks after injury

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196